CLINICAL TRIAL: NCT01039103
Title: A Randomized, International, Multi Centre Study to Assess the Efficacy and Safety of Intravenous PEG-liposomal Prednisolone Sodium Phosphate (Nanocort®) vs Intravenous Methylprednisolone (Solu-Medrol®) Treatment in Patients With Acute Exacerbation of Relapsing-remitting Multiple Sclerosis or in Patients With Clinically Isolated Syndrome (CIS)
Brief Title: Nanocort in Acute Exacerbation of Relapsing-Remitting Multiple Sclerosis (MS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: GLPG0303-CL-204; 2009-013884-21 (EudraCT Number)
Record Dates: First submitted 2009-12-20; First posted 2009-12-24 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Acute Exacerbation of Remitting Relapsing Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: PEG-liposomal prednisolone sodium phosphate
MeSH Terms: interventions — Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nanocort (Experimental): PEG-liposomal prednisolone sodium phosphate (Nanocort) 300 mg intravenous (IV), single dose 500 ml infusion over at least 2 hours on day 1
  Interventions: Drug: PEG-liposomal prednisolone sodium phosphate
- Solu-Medrol (Active Comparator): Methylprednisolone (Solu-Medrol) 1 g, IV, infusion over 2 hours on days 1, 2 and 3
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: PEG-liposomal prednisolone sodium phosphate — PEG-liposomal prednisolone sodium phosphate 300 mg intravenous (IV), single dose 500 ml infusion over at least 2 hours on day 1
  Other Names: Nanocort
  Arms: Nanocort
Drug: Methylprednisolone — Methylprednisolone 1 g, IV, infusion over 2 hours on days 1, 2 and 3
  Other Names: Solu-Medrol
  Arms: Solu-Medrol

SUMMARY:
Patients with an acute exacerbation of Relapsing-Remitting Multiple Sclerosis or with Clinically Isolated Syndrome receive either one single infusion of Nanocort or three daily infusions of SoluMedrol. Main objective is to assess the occurrence of new gadolinium-enhanced T1-weighted lesions at week 8 vs week 1 after treatment.

ELIGIBILITY:
INCLUSION criteria

* Diagnosis of RRMS (per McDonald criteria, 2005) with dissemination in time and space OR a diagnosis of CIS confirmed by MRI. Patients with CIS who only have optic neuritis will be excluded from this study
* A maximum Expanded Disability Status Scale (EDSS) score of ≤ 6
* New neurological symptoms or exacerbation of prior neurological symptoms of over 24 hours duration but <7 days duration, verified by neurological examination

EXCLUSION criteria:

* Primary progressive MS.
* Secondary progressive MS without superimposed relapses.
* Received systemic corticosteroids within 4 weeks of screening for treatment of MS or other conditions.
* any contraindication for treatment with (systemic) corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in gadolinium-enhanced T1-weighted lesions according to the McDonald criteria (2005) from Day 8 to Week 8. | 8 weeks

SECONDARY OUTCOMES:
Change in gadolinium-enhanced T1-weighted lesions according to the McDonald criteria (2005) from Day 8 to Week 4. | 4 weeks
Quality of life measured by changes in MSIS-29 | 12 weeks
Clinical response measured by changes in MSFC | 12 weeks
Plasma levels of free prednisolone and prednisolone phosphate | 12 weeks
Occurrence of adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johan Beetens, PhD, Study Director — Galapagos NV
Locations (8):
- Belgium (3):
  - Departement Neurologie AZ St Jan AV, Bruges
  - Nationaal MS Centrum, Melsbroek
  - Revalidatie & MS-centrum Overpelt, Overpelt
- Germany (3):
  - Krankenhaus Hohe Warte, Neurologische Klinik, Bayreuth
  - St. Josef Hospital der Ruhr, Bochum
  - Klinikum Rechts der Isar der technischen Universitaet Muenchen, Neurologische Klinik und Poliklinik, München
- Poland (2):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Diagnomed-Clinical Research Sp. z o.o., Katowice